CLINICAL TRIAL: NCT06454357
Title: A Phase II/III Clinical Study to Evaluate the Efficacy and Safety of B007 in Subjects With Pemphigus.
Brief Title: A Clinical Study of B007 in the Treatment of Pemphigus.
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shanghai Jiaolian Drug Research and Development Co., Ltd (Industry)
Collaborators: Shanghai Pharmaceuticals Holding Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPH-B007-304
Record Dates: First submitted 2024-06-06; First posted 2024-06-12 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-06

CONDITIONS: Pemphigus
MeSH Terms: conditions — Pemphigus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- B007 (Experimental)
  Interventions: Drug: B007

INTERVENTIONS:
Drug: B007 — B007：high dose/low dose: Subcutaneous injection was administered on days 1 and 15

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of B007 in subjects with pemphigus.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who voluntarily participate in this study and sign informed consent form;
2. Subjects who meet the clinical manifestations of pemphigus and are clinically diagnosed as prescribed diseases;
3. Subjects with first diagnosis or relapse;
4. Subjects who have the ability to follow the study protocol as determined by the investigator.

Exclusion Criteria:

1. Subjects diagnosed with prescribed diseases;
2. Since the diagnosis of pemphigus, Disease duration>4 years;
3. Subjects using prescribed drugs;
4. Presence of a specified disease or history of disease;
5. The subjects has prescribed examination abnormalities that are assessed as unsuitable for participation in the study by the investigator;
6. A history of severe allergy or allergic reaction to human or mouse monoclonal antibodies; known contraindications to orally prescribed drugs;
7. Subjects who participate in another interventional clinical trial at a specified time before randomization;
8. Subjects who received live vaccine at the specified time before the first dose and are expected to receive the vaccine at the specified time after the last dose;
9. Pregnant and lactating women;
10. Fertile female subjects do not agree to use effective contraception from signing the informed consent form to the prescribed time after the last dose.

    Women who are considered fertile by the investigator must have negative serum pregnancy tests before starting the drug;
11. Sexually active male subjects who do not intend to use an effective contraceptive method during the trial period or within specified time after the last dose, or male subjects who plan to donate sperm at a specified time during the trial or after the last dose.
12. Other conditions deemed unsuitable for participation in this study by the researchers.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2024-07-12 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects：Complete remission with minimal treatment | Approximately36 weeks

SECONDARY OUTCOMES:
The number of relapses of the disease | Approximately 1 years
Proportion of subjects：Partial remission | Approximately 36weeks
Change: PDAI（Pemphigus disease area index） | Approximately 36 weeks
CR/PR Proportion of subjects：Complete remission /Partial remission | Approximately 52 weeks
DoR （Duration of Response） | Approximately 1 years
Incidence of Treatment-Emergent Adverse Events | Approximately 1 years

CONTACTS AND LOCATIONS:
Locations (12):
- China (12):
  - Peking University First Hospital, Beijing
  - The Second Xiangya Hospital of Central South University, Changsha
  - Chengdu Second People's Hospital, Chengdu
  - West China Hospital, Sichuan University, Chengdu
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou
  - Dermatology Hospital of Southern Medical University, Guangzhou
  - Guangdong Provincial People's Hospital, Guangzhou
  - Shandong First Medical University-Affiliated Skin Hospital, Jinan
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan
  - Henan Provincial People's Hospital, Zhengzhou